CLINICAL TRIAL: NCT06092268
Title: A Phase IB/II, Open-Label, Multicentre Clinical Study to Evaluate the Safety, Tolerability and Efficacy of SHR-A2009 for Injection in Combination With Other Therapies in Patients With Advanced Solid Tumors
Brief Title: A Phase IB/II Clinical Study of SHR-A2009 for Injection in Combination With Other Antitumor Therapies in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A2009-201
Record Dates: First submitted 2023-10-08; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Part A: SHR-A2009 for injection in combination with Almonertinib Mesilate Tablets (Experimental)
  Interventions: Drug: SHR-A2009 for injection ； Almonertinib Mesilate Tablets
- Treatment Part B: SHR-A2009 for injection in combination with Adebrelimab Injection (Experimental)
  Interventions: Drug: SHR-A2009 for injection；Adebrelimab Injection

INTERVENTIONS:
Drug: SHR-A2009 for injection ； Almonertinib Mesilate Tablets — Phase IB: SHR-A2009 will be administered intravenously，Almonertinib Mesilate Tablets will be administered orally. 2 or 3 dose levels are preset in phase IB.
  Phase II: 2 dose cohorts will be selected and it's randomization.
  Arms: Treatment Part A: SHR-A2009 for injection in combination with Almonertinib Mesilate Tablets
Drug: SHR-A2009 for injection；Adebrelimab Injection — Phase IB: SHR-A2009 and Adebrelimab will be administered intravenously. 2 dose levels are preset in phase IB.
  Phase II: RPD2 will be selected to evaluate preliminary efficacy.
  Arms: Treatment Part B: SHR-A2009 for injection in combination with Adebrelimab Injection

SUMMARY:
This study is an open-label, multicenter Phase IB/II clinical trial to evaluate the safety, tolerability, pharmacokinetics and efficacy of SHR-A2009 for injection in combination with other antitumor therapies in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 75 years old (inclusive), Female or male
2. Subjects with unresectable locally advanced or metastatic non-small cell lung cancer confirmed by histology or cytology
3. Previously treated by EGFR-TKI or other standard treatment or have not been treated for metastatic setting;
4. At least one measurable tumor lesion according to RECIST v1.1 (enrollment of subjects with only non-target lesions is permitted in Stage IB phase)
5. ECOG performance score of 0-1;
6. Expected survival time ≥ 12 weeks;
7. Adequate bone marrow and organ function
8. Subjects are required to give informed consent for this study prior to the trial and voluntarily sign a written informed consent form.

Exclusion Criteria:

1. Subjects with active central nervous system (CNS) metastases.
2. Spinal cord compression not cured by surgery and/or radiotherapy cannot be enrolled.
3. Subjects with uncontrolled tumor-related pain
4. Clinically uncontrollable third space fluid
5. Received antitumor therapy such as chemotherapy within 4 weeks prior to the first dose of study drug;
6. Received >30 Gy of non-thoracic radical radiation therapy within 4 weeks prior to the first administration of study drug;
7. Major organ surgery or significant trauma within 4 weeks prior to first use of study drug;
8. Concomitant other malignancies ≤ 5 years prior to first dose of study drug;
9. Subjects with a history of interstitial pneumonitis or imaging at screening suggestive of suspected interstitial pneumonitis; or other moderate-to-severe lung disease that severely affects lung function
10. Serious cardiovascular disease
11. Presence of refractory nausea, vomiting, chronic gastrointestinal disease, etc.; subjects with active, known or suspected autoimmune diseases
12. Presence of severe infection within 4 weeks prior to first dose of study drug
13. Subjects with clinically significant bleeding symptoms within 3 months prior to the first dose of study drug
14. Arterial/venous thrombotic events within 3 months prior to the first study dose
15. History of immunodeficiency, including a positive HIV test
16. Presence of active hepatitis B or C;
17. History of severe allergic reactions to other monoclonal antibodies or allergic reactions to any component of the SHR-A2009 product.
18. Known history of alcohol or drug dependence or addiction;
19. Persons with mental disorders or poor compliance;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity (DLT) (phase IB) | 21 days after the first dose was administered to each subject.
Objective Response Rate (ORR) (phase II). | 2 years

SECONDARY OUTCOMES:
PK parameter: toxin-binding antibody of SHR-A2009 | through study completion, an average of 2 years
PK parameter: total antibody of SHR-A2009 | through study completion, an average of 2 years
PK parameter: free toxin of SHR-A2009 | through study completion, an average of 2 years
Plasma concentration of Adebrelimab | through study completion, an average of 2 years
Immunogenicity of SHR-A2009 and Adebrelimab (Anti-SHR-A2009 antibody, anti- Adebrelimab antibody ) (Phase IB) | through study completion, an average of 2 years
Duration of response(DoR ) | One year after the last subject was enrolled in the group
Progression Free Survival(PFS) | 2 years after the last subject was enrolled in the group
Objective response rate | 2 years after the last subject was enrolled in the group
overall survival (OS) (phase IB) | 3 years after the last subject was enrolled in the group
Incidence of AEs（Phase II (efficacy expansion phase)） | from Day1 to 90 days after last dose
Incidence of SAEs（Phase II (efficacy expansion phase)） | from Day1 to 90 days after last dose

IPD SHARING:
Plan to Share IPD: Undecided